CLINICAL TRIAL: NCT05741619
Title: Long-term Follow up of Patient With Anti-GABAbr Antibodies Associated-encephalitis.
Acronym: SALTEA GABAbr
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 897
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Autoimmune Encephalitis
Keywords: anti-GABAbr; autoimmune encephalitis; outcome
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Sera and CSF at the diagnosis have been stocked in biobank (samples are already stored in biobank repositories and collected as part of "good clinical practice")
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-GABABr encephalitis: This is a non-interventional study involving clinical data. This data are information of medical follow up on patient like diagnosis, symptoms, biological results, cancer, treatments.
  Interventions: Other: Long-term outcome

INTERVENTIONS:
Other: Long-term outcome — Autonomy, physical examination, behavioural disorders

SUMMARY:
First described in 2010, GABA-B-receptor antibodies-associated encephalitis is a disease with a severe vital and functional prognosis. Indeed, functional status is mostly altered by encephalitis and it induced consequences while vital status is mostly engaged by cancer very often associated in the course of the disease, mostly small-cell lung cancer (SCLC).

While knowledge is growing on clinical features at each stage of the disease, long-term outcome data is still lacking even if known to be pejorative.

In this study, we aimed to describe long-term follow up of all patients who were diagnosed a GABAb-receptor antibodies-associated encephalitis in the French Paraneoplastic Neurological Syndrome Reference Center until now.

ELIGIBILITY:
Inclusion Criteria:

* encephalitis tested positive to GABAbr-antibodies after the examination of CSF samples tested for autoimmune encephalitis at the French Paraneoplastic Neurological Syndrome Reference Center from January 2011 to January 2022.

Exclusion Criteria:

* tested positive to another onconeural antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of reference center on paraneoplastic neurological syndrom
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Modified-Rankin scale (mRS) | At 60 month (after the beginning of the disease)
  Modified-Rankin scale (mRS) ranked from 0 (full autonomy) to 6 (death)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon, France